CLINICAL TRIAL: NCT01857700
Title: Compensation for Transport Costs and Lost Wages Associated With Voluntary Medical Male Circumcision (VMMC) Uptake: an Intervention to Increase VMMC Demand Among Older Men in Nyanza Province
Brief Title: Economic Compensation to Increase Demand for Voluntary Medical Male Circumcision
Acronym: CTT-VMMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Impact Research & Development Organization (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 12-1961
Record Dates: First submitted 2013-05-07; First posted 2013-05-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Voluntary Medical Male Circumcision; Circumcision Adult
MeSH Terms: interventions — Compensation and Redress; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conditional economic compensation (Experimental): A scratch off card will be used to randomly determine which of the compensations will be offered: compensation for transport cost, compensation for lost wages, or compensation for transport cost and lost wages
  Interventions: Other: Compensation for transport cost; Other: Compensation for lost wages; Other: Compensation for transport cost and lost wages
- Standard of Care (Placebo Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Compensation for transport cost
  Arms: Conditional economic compensation
Other: Compensation for lost wages
  Arms: Conditional economic compensation
Other: Compensation for transport cost and lost wages
  Arms: Conditional economic compensation
Other: Standard of Care — Consistent with standard of care, participants in this group will be offered a refreshment during their office visit.
  Arms: Standard of Care

SUMMARY:
Research questions: What effect does provision of food vouchers have on uptake of voluntary medical male circumcision? What is the amount of food voucher that should be given?

Hypothesis: The percentage of men who are compensated for costs of travel to and lost wages due to VMMC and who undergo VMMC will be higher than the percentage of men who are compensated for lost wages or travel and undergo VMMC, and both of these percentages will be higher than the percentage of men who are not compensated for travel or lost wage costs but undergo VMMC.

DETAILED DESCRIPTION:
Purpose: Implement a randomized trial to test whether offering compensation to older men conditional on their coming for medical male circumcision can increase uptake of circumcision services.

Participants: 1,500 uncircumcised men of ages 25-49 in Nyando District, 21 men who chose to be circumcised and 21 who did not get circumcised, 10 female partners of men who became circumcised and 10 female partners of men who did not will be interviewed

Procedures (methods): To increase uptake of male circumcision, investigators will offer conditional economic compensation for male circumcision. Randomly selected study participants will be given the opportunity, conditional on undergoing male circumcision, to obtain food vouchers that are intended to offset the cost of accessing the VMMC services and the potential lost work the day of the procedure and in the 2 days following the procedure. The food vouchers will be given after study participants choose to uptake VMMC services at any of the static or outreach sites operated by Impact Research and Development Organization (IRDO). Participants will be randomized to one of three intervention groups or to a control group. Participants in the intervention groups will have the opportunity to receive a food voucher valued at one of three amounts (in KES, Kenyan Shillings) if they choose to get circumcised. Participants in the control group will receive a soda but no food voucher if they choose to get circumcised. The amounts for the intervention groups were selected based on the approximate value of 3 days of work and average transportation costs within the district. The amounts were also chosen so that they are not so large as to be perceived as coercive. Investigators selected food vouchers instead of cash or mobile phone credit because the vouchers were deemed to be more acceptable given the sensitive nature of the intervention and men's concern with feeding their families; it was also considered more logistically feasible to offer vouchers at the health facilities rather than cash. Additional focus group discussions will be held to verify that this form and amount of compensation is acceptable and desirable in study communities and if necessary, the intervention can be changed based on these results.

The food vouchers will be valid at dukas (shops) located within the district. At the beginning of the study, these shops will be visited and informed about ways to receive cash for the vouchers at the central IRDO office in Nyando District. IRDO has previously explored the feasibility of implementing the voucher scheme and found that it can be implemented in the study areas.

Three months after enrollment of study participants, investigators will conduct qualitative research in which there will be in-depth interviews with a small sample of men who did and did not come for circumcision and with their partners. Three topics will be examined in the qualitative interview: men's decision-making, logistics of the intervention, and women's perceptions.

ELIGIBILITY:
Inclusion Criteria:

Men

* aged 25-49
* living in enumerated locations and sublocations of Nyanza Province
* who intend to remain in their village for the next three months.

Female partners of some of these eligible men are also eligible to be interviewed about their perceptions.

Exclusion Criteria:

Men

* younger than 25,
* older than 49, or
* intending to move away from their village within three months.

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1504 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
percentage who undergo voluntary medical male circumcision | 14 weeks

SECONDARY OUTCOMES:
Qualitative Outcome Measure #1: men's decision-making around circumcision, including how the food voucher affected their decision and communications with their female partners surrounding circumcision. | 14 weeks
  men's concerns with circumcision (i.e., what man had heard about circumcision prior to enrollment; what man had thought about getting circumcised prior to enrollment; greatest concern with getting circumcised prior to enrollment; degree of financial barrier prior to enrollment), experience with how food voucher was explained (i.e., what man was told about voucher amount, what man was told about reason for voucher, what man was told about how it could be redeemed, whether anything was unclear, whether questions were answered satisfactorily), what was discussed with a female partner (i.e., whether circumcision had ever been discussed; her opinion of it; whether the study and food voucher were discussed and what was discussed; her opinion of the study and food voucher; her opinion of whether man should get circumcision; whether partner's opinions influenced man's decision about whether to go for circumcision)
Qualitative Outcome Measure #2: impact of food voucher intervention on man | 14 weeks
  the effect of the food voucher on the man (i.e., whether it was volunteered as the biggest reason for deciding to get circumcised; whether it had changed his mind about getting circumcised; whether the value of the food voucher made it easier or more difficult to decide about getting circumcised)
Qualitative Outcome Measure #3: impact of intervention logistics on man | 14 weeks
  use of food voucher (i.e., whether redeeming it with 30 days was a constraint; whether there were any problems with redeeming it) and transportation & time away from work (i.e., distance between residence and nearest circumcision clinic; transportation to clinic and its total cost, number of days missed from work and lost wages because of missed work; whether the food voucher offset the costs of transportation and lost wages).

OTHER OUTCOMES:
Qualitative Outcome Measure #4: couple's decision-making around circumcision (including how the food voucher affected their decision and communications with male partners surrounding circumcision) as reported by female partner | 14 weeks
  woman's concerns with circumcision (i.e., what woman had heard about circumcision prior to partner's enrollment; what woman had thought about getting circumcised prior to partner's enrollment; greatest concern with partner getting circumcised prior to his enrollment; degree of financial barrier prior to enrollment), experience with how food voucher was explained (i.e., what woman was told about voucher amount, what woman was told about reason for voucher, what woman was told about how it could be redeemed, whether anything was unclear, whether questions were answered satisfactorily), what was discussed with a partner (i.e., whether circumcision had ever been discussed; her opinion of it; whether the study and food voucher were discussed and what was discussed; partner's opinion of the study and food voucher; his opinion of whether he should get circumcision; whether her opinions influenced man's decision about whether to go for circumcision)
Qualitative Outcome Measure #5: impact of food voucher intervention on couple, as reported by female partner | 14 weeks
  the effect of the food voucher on the couple (i.e., whether it was volunteered as the biggest reason for deciding that man would get circumcised; whether it had changed couple's mind about getting circumcised; whether the value of the food voucher made it easier or more difficult for couple to decide about getting circumcised)
Qualitative Outcome Measure #6: impact of intervention logistics on couple, as reported by female partner | 14 weeks
  use of food voucher (i.e., whether redeeming it with 30 days was a constraint for the couple; whether there were any problems for the couple with redeeming it) and transportation & time away from work (i.e., distance between residence and nearest circumcision clinic; transportation to clinic and its total cost, number of days missed from work and lost wages because of missed work; whether the food voucher offset the costs of transportation and lost wages).

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — UNC-Chapel Hill, CPC and SPH-HPM
Locations (1):
- Impact Research & Development Organization, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Thirumurthy H, Masters SH, Rao S, Bronson MA, Lanham M, Omanga E, Evens E, Agot K. Effect of providing conditional economic compensation on uptake of voluntary medical male circumcision in Kenya: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):703-11. doi: 10.1001/jama.2014.9087. PMID 25042290
- See also: This study is funded by the Bill & Melinda Gates Foundation. — http://www.gatesfoundation.org/